CLINICAL TRIAL: NCT02622100
Title: Evaluation of Effectiveness and Safety of Bioresorbable Vascular Scaffold in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: Evaluation of Effectiveness and Safety of Bioresorbable Vascular Scaffold in Routine Clinical Practice
Acronym: IRIS BVS
Status: Terminated | Type: Observational
Why Stopped: Due to stop BVS supply discontinuation
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Principal investigator, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2015-11
Record Dates: First submitted 2015-11-29; First posted 2015-12-04 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Arterial Occlusive Diseases; Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease
Keywords: Bioresorbable Vascular Scaffold; Routine Clinical Practice; Angioplasty, Transluminal, Percutaneous Coronary; Coronary Artery Disease; drug eluting stent
MeSH Terms: conditions — Arterial Occlusive Diseases; Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bioresorbable Vascular Scaffold
  Interventions: Device: Bioresorbable Vascular Scaffold

INTERVENTIONS:
Device: Bioresorbable Vascular Scaffold

SUMMARY:
The purpose of this study is to evaluate the relative effectiveness and safety of Bioresorbable Vascular Scaffold compared to other (drug eluting stents) DES.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Intervention with Bioresorbable Vascular Scaffold
* Agreed with written informed consent form

Exclusion Criteria:

* Bypass graft surgery (CABG) recommended
* Lesion with previous bypass graft surgery (CABG)
* Severe calcification and/or severe tortuosity
* Contraindication to antiplatelet agent or Inability to take dual antiplatelet therapy within 1 year
* Life expectancy of 1year and under
* Subjects scheduled to receive cardiac surgery or serious non-cardiac surgery
* Cardiac shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Bioresorbable Vascular Scaffold
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Composite event | 1 year
  The number of events with the first occurrence of a composite event(death, non-fatal myocardial infarction, target vessel revascularization)

SECONDARY OUTCOMES:
all death | 5 years
cardiac death | 5 years
myocardial infarction | 5 years
Composite event of death or myocardial infarction | 5 years
Composite event of cardiac death or myocardial infarction | 5 years
Target Vessel revascularization | 5 years
  Defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion, which includes upstream and downstream branches and the target lesion itself.
  Clinical-driven Clinically indicated angiography at follow-up shows a percent diameter stenosis ≥ 50% (core lab QCA assessment) and if one of the following occurs: (1) a positive history of recurrent angina pectoris, presumably related to the target vessel; (2) objective signs of ischemia at rest (ECG changes) of during exercise test (or equivalent), presumably related to the target vessel; (3) abnormal results of any invasive functional diagnostic test (eg, Doppler flow velocity reserve, fractional flow reserve).
  Ischemia-driven if one of followings of above-mentioned symptom (clinical-driven) or sign of ischemia or diameter stenosis ≥ 70 %
Target Lesion revascularization | 5 years
  Defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLRs should be classified prospectively as clinically indicated or not clinically indicated by the investigator prior to repeat angiography. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement. The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the stent.
Stent thrombosis | 5 years
  DEFINITE stent thrombosis : acute coronary syndrome and angiographic or pathologic evidence of stent thrombosis; PROBABLE stent thrombosis : unexplained death within 30 days or target-vessel infarction without angiographic information Academic Research Consortium (ARC) stent thrombosis is reported as a cumulative value at different time points and within the different separate time points. Time 0 is the time point after the guide catheter has been removed. Acute stent thrombosis: 0-24 hours after stent implantation; Subacute stent thrombosis: >24 hours to 30 days post; late stent thrombosis: >30 days to 1 year post; Very late stent thrombosis: >1 year post;
Stroke | 5 years
Procedural success | 3 days
  Defined as mean lesion diameter stenosis ≤50% and without the occurrence of in-hospital myocardial infarction (MI), target vessel revascularization (TVR), or death

CONTACTS AND LOCATIONS:
Locations (14):
- South Korea (14):
  - Asan Medical Center, Seoul, Songpa-gu
  - Hallym University Sacred Heart Hospital, Anyang
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - ChonBuk National University Hospital, Jeonju
  - Bundang CHA Hospital, Seongnam
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hosp, Wŏnju

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.